CLINICAL TRIAL: NCT05923346
Title: Educational Intervention on Celiac Disease and Gluten-free Diet Through Social Networks (GLUTLEARN Project).
Acronym: GLUTLEARN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Itziar Churruca Ortega, Profesor Titular de Universidad - University Tenured Professor, University of the Basque Country (UPV/EHU)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: M10_2020_081 GLUTLEARN; GIU18/78 (Other Grant/Funding Number: University of the Basque Country (UPV/EHU)); GIU21/053 (Other Grant/Funding Number: University of the Basque Country (UPV/EHU)); IT-1419-19 (Other Grant/Funding Number: Basque Government); University-Society US22/22 (Other Grant/Funding Number: University of the Basque Country (UPV/EHU))
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Celiac Disease
Keywords: celiac disease; nutrition education; gluten-free diet; balanced diet; social networks
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glutlearn (Experimental)
  Interventions: Other: GLUTLEARN

INTERVENTIONS:
Other: GLUTLEARN — The group will be made up of users of the social network Instagram who have celiac disease or are close to a celiac patient (parent/guardian of celiac children or cohabitants).
  The intervention will be carried out through the social network Instagram. Participants will be recruited through the same social network. Participants must agree to take part in the study.
  The educational intervention will be carried out for one month, where each day a "post" will be uploaded with specific, truthful and current information. The content of the intervention has been divided into 5 main blocks: 1) general concepts about CD, 2) balanced GFD, 3) food labelling, 4) cross-contact/cross-contamination, 5) new research on CD and useful resources for disease management.

SUMMARY:
Celiac disease (CD) is an autoimmune disease that occurs in people who are genetically predisposed to gluten consumption (1). The prevalence of the disease is about 1-2% and it is more common in women than in men, and in children than in adults (2).

The only current treatment for celiac disease is a strict, lifelong gluten-free diet. This involves the complete elimination of gluten from the diet. Gluten is not only present in some cereals such as wheat, rye, barley and oats, but is also found in many foods that have been processed. In addition to being safe, the gluten-free diet must also be balanced.

Following a gluten-free diet creates psychological and social problems for the people who have to follow it (3). It has been seen in several studies that people with celiac condition can feel different and excluded, as it is difficult to eat out, to make sure that the food is gluten-free and to avoid cross-contact (4-8).

Due to the complicate situation of people with celiac disease, they do not hesitate to seek information about the management of their diseas. That is why people with celiac disease turn to social networks, as a rapid, visual and accessible way to share information (9-11).

In line with the objectives of the University to which the Gluten3S research group belongs to (University of the Basque Country, UPV/EHU), the group has been aware for some time of the importance of disseminating science on social networks in order to make the results of the research reach the general public. It is considered that creating a nutritional education programme about CD and Gluten-Free Diet (GFD), delivered by experts in the field, could be useful in improving knowledge and attitudes about this matter. This will empower people with CD to improve their self-care and take control of their situation. Furthermore, it is also interesting to design the programme in such a way that the impact of the intervention can be measured, always with the intention of continuous improvement and reaching people with celiac disease and their environment in an effective way.

The educational intervention will be carried out for one month and is aimed at adults with coeliac disease or adults with coeliac relatives who are involved in their care. Each day a post will be uploaded to Instagram with specific, accurate and current information. The content of the intervention has been divided into 5 main blocks: 1) general concepts about CD, 2) balanced GFD, 3) food labelling, 4) cross-contact/cross-contamination, 5) new research on CD and useful resources for disease management.

The evaluation of the intervention will be carried out through pre- and post-intervention questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age
* Have celiac disease or be involved in the care of a person with celiac disease
* Be an Instagram user

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Knowledge regarding celiac disease | 5 weeks
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test) in order to assess changes due to the intervention.The unit of measure will be the score obtained in the questionnaires (0, worst-1,best/0, disagree-4,agree/the number of correct answers).
Attitude towards celiac disease: degree of concern | 5 weeks
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test) in order to assess changes due to the intervention.The unit of measure will be the score obtained in the questionnaires (0, worst-1,best/0, disagree-4,agree/the number of correct answers).
Knowledge regarding balanced GFD | 5 weeks
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test) in order to assess changes due to the intervention.The unit of measure will be the score obtained in the questionnaires (0, worst-1,best/0, disagree-4,agree/the number of correct answers).
Knowledge regarding food labels | 5 weeks
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test) in order to assess changes due to the intervention.The unit of measure will be the score obtained in the questionnaires (0, worst-1,best/0, disagree-4,agree/the number of correct answers).
Attitude: degree of confidence in their choice of food | 5 weeks
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test) in order to assess changes due to the intervention.The unit of measure will be the score obtained in the questionnaires (0, worst-1,best/0, disagree-4,agree/the number of correct answers).
Knowledge regarding cross-contact | 5 weeks
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test) in order to assess changes due to the intervention.The unit of measure will be the score obtained in the questionnaires (0, worst-1,best/0, disagree-4,agree/the number of correct answers).
Attitude: degree of confidence in avoiding cross-contact | 5 weeks
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test) in order to assess changes due to the intervention.The unit of measure will be the score obtained in the questionnaires (0, worst-1,best/0, disagree-4,agree/the number of correct answers).
Knowledge regarding new research in CD | 5 weeks
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test) in order to assess changes due to the intervention.The unit of measure will be the score obtained in the questionnaires (0, worst-1,best/0, disagree-4,agree/the number of correct answers).

SECONDARY OUTCOMES:
Satisfaction about the education received | Immediately after the intervention
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test). Secondary outcomes will be measured in the post-questionnaire. • The unit of measure will be the score obtained in the questionnaires (0, disagree-4,agree).
Perception of the importance of educational activities | Immediately after the intervention
  A questionnaire will be used to be able to assess all outcomes. The same questionnaire will be completed twice, once before the intervention (pre-test) and again immediately after the end of the intervention (post-test). Secondary outcomes will be measured in the post-questionnaire. • The unit of measure will be the score obtained in the questionnaires (0, disagree-4,agree).

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Basque Country (UPV/EHU), Vitoria-Gasteiz, Álava, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebwohl B, Rubio-Tapia A. Epidemiology, Presentation, and Diagnosis of Celiac Disease. Gastroenterology. 2021 Jan;160(1):63-75. doi: 10.1053/j.gastro.2020.06.098. Epub 2020 Sep 18. PMID 32950520
- [Background] Singh P, Arora A, Strand TA, Leffler DA, Catassi C, Green PH, Kelly CP, Ahuja V, Makharia GK. Global Prevalence of Celiac Disease: Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2018 Jun;16(6):823-836.e2. doi: 10.1016/j.cgh.2017.06.037. Epub 2018 Mar 16. PMID 29551598
- [Background] Itzlinger A, Branchi F, Elli L, Schumann M. Gluten-Free Diet in Celiac Disease-Forever and for All? Nutrients. 2018 Nov 18;10(11):1796. doi: 10.3390/nu10111796. PMID 30453686
- [Background] Rosen A, Ivarsson A, Nordyke K, Karlsson E, Carlsson A, Danielsson L, Hogberg L, Emmelin M. Balancing health benefits and social sacrifices: a qualitative study of how screening-detected celiac disease impacts adolescents' quality of life. BMC Pediatr. 2011 May 10;11:32. doi: 10.1186/1471-2431-11-32. PMID 21569235
- [Background] Olsson C, Lyon P, Hornell A, Ivarsson A, Sydner YM. Food that makes you different: the stigma experienced by adolescents with celiac disease. Qual Health Res. 2009 Jul;19(7):976-84. doi: 10.1177/1049732309338722. PMID 19556403
- [Background] Cadenhead JW, Wolf RL, Lebwohl B, Lee AR, Zybert P, Reilly NR, Schebendach J, Satherley R, Green PHR. Diminished quality of life among adolescents with coeliac disease using maladaptive eating behaviours to manage a gluten-free diet: a cross-sectional, mixed-methods study. J Hum Nutr Diet. 2019 Jun;32(3):311-320. doi: 10.1111/jhn.12638. Epub 2019 Mar 5. PMID 30834587
- [Background] Wolf RL, Lebwohl B, Lee AR, Zybert P, Reilly NR, Cadenhead J, Amengual C, Green PHR. Hypervigilance to a Gluten-Free Diet and Decreased Quality of Life in Teenagers and Adults with Celiac Disease. Dig Dis Sci. 2018 Jun;63(6):1438-1448. doi: 10.1007/s10620-018-4936-4. Epub 2018 Jan 31. PMID 29387990
- [Background] Singh P, Dennis M. Eliminating Dietary Gluten: Don't Be a "Glutton for Punishment". Dig Dis Sci. 2018 Jun;63(6):1374-1375. doi: 10.1007/s10620-018-5010-y. No abstract available. PMID 29546643
- [Background] Al Sarkhy A. Social media usage pattern and its influencing factors among celiac patients and their families. Saudi J Gastroenterol. 2020 Mar-Apr;26(2):99-104. doi: 10.4103/sjg.SJG_495_19. PMID 32031161
- [Background] McNally SL, Donohue MC, Newton KP, Ogletree SP, Conner KK, Ingegneri SE, Kagnoff MF. Can consumers trust web-based information about celiac disease? Accuracy, comprehensiveness, transparency, and readability of information on the internet. Interact J Med Res. 2012 Apr 4;1(1):e1. doi: 10.2196/ijmr.2010. PMID 23611901
- [Background] Trovato CM, Montuori M, Oliva S, Cucchiara S, Cignarelli A, Sansone A. Assessment of public perceptions and concerns of celiac disease: A Twitter-based sentiment analysis study. Dig Liver Dis. 2020 Apr;52(4):464-466. doi: 10.1016/j.dld.2020.02.004. Epub 2020 Feb 29. No abstract available. PMID 32127326
- [Result] Vazquez-Polo M, Navarro V, Larretxi I, Perez-Junkera G, Lasa A, Matias S, Simon E, Churruca I. Uncovering the Concerns and Needs of Individuals with Celiac Disease: A Cross-Sectional Study. Nutrients. 2023 Aug 22;15(17):3681. doi: 10.3390/nu15173681. PMID 37686713